CLINICAL TRIAL: NCT03217903
Title: High Risk Myelodysplasia Treated by Azacytidine : Genetic and Epigenetic (MYRAGE)
Acronym: MYRAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Inserm U954 - N-GERE (Nutrition, Genetics and Exposition to Environmental Risk) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MYRAGE
Record Dates: First submitted 2017-07-03; First posted 2017-07-14 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: High-risk Myelodysplastic Syndromes With Excess Blasts
Keywords: Myelodysplastic syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Myelography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with High-risk MDS With Excess Blasts (Experimental)
  Interventions: Diagnostic Test: Myelogram

INTERVENTIONS:
Diagnostic Test: Myelogram — Bone marrow aspiration after 3 cycles of Azacytidine treatment

SUMMARY:
Myelodysplastic syndromes (MDS) are the most frequent myeloid neoplasms in Western Countries.They mainly affect patients aged 65 years or older. This is a very heterogenous group of diseases, which prognosis is evaluated with International Prognosis Scoring System. High risk MDS present with high frequency of transformation into acute myeloid leukemia. Treatment of high risk MDS often is based on hypomethylating agents, such as 5'-azacytidine (Azacytidine), with a complete response in approximativel 20% of cases..

This treatment is based on 4-week cycles, with daily injection during the first week and rest during the 3 next weeks of the cycle.

Azacytidine efficacy is commonly evaluated with clinical and biological parameters determined by the International Working Group 2006. These parameters are usually evaluated after at least 6 cycles of treatments.

There is a response with Azacytidine treatment in 60% of cases, including 40% of partial responses and 20% of complete responses. In 40% of patients, there is no response, which means that the disases is stable or in progression under therapy.

In this regard, early evaluation of treatment response is an issue. We want to improve our knowledge about early response criteria in Azacytidine-treated high-risk MDS, focusing on SMD with excess blasts, which represent 30 to 40% of total MDS.

Then, the investigator team want to compare DNA methylation profile at diagnosis and after 3 cycles of Azacytidine treatment.

Main objective :

Identify DNA methylation profiles related to response to Azacytidine therapy, after only 3 cycles of treatment, in high risk MDS with excess blasts.

Secondary objective :

Identify at diagnosis DNA methylation profiles that are predicitive of response to Azacytidin, in high risk MDS with excess blasts.

ELIGIBILITY:
Pre-inclusion Criteria:

* patient benefiting from social welfcare
* patient followed at the University Hospital of Nancy
* patient aged 18 years or older
* patient informed on research organization and having signed an informed pre-inclusion consent
* No personal history of myelodysplastic syndrome
* clinical exam adapted to research
* one or more blood cytopenia

Inclusion Criteria:

* patient benefiting from social welfcare
* patient followed at the University Hospital of Nancy
* patient aged 18 years or older
* patient informed on research organization and having signed an informed inclusion consent
* definitive diagnosis of high risk myelodysplastic syndrome with excess blasts
* eligibility to an Azacytidine therapy as first-line treatment

Exclusion Criteria:

* personal history or current other cancer
* immediate acute myeloid leukemia
* personal history of demethylation treatment
* pregnant or breast feeding women
* life-theatening condition
* guardianship
* imprisoned patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Methylation level of the Differentially Methylated Regions (DMR) | 3 months (after 3 cycles of treatment)
Overall response by IWG 2006 response criteria (complete remission / partial remission / non response) | At the treatment response assessment (After 6-12 cycles of treatment up to 52 weeks)

SECONDARY OUTCOMES:
Methylation level of the Differentially Methylated Regions (DMR) | At diagnosis
Cytogenetic response by IWG 2006 response criteria (major / minor / no response) | At the treatment response assessment (After 6-12 cycles of treatment up to 52 weeks)
Hematologic improvement by IWG 2006 response criteria (major / minor / no response) | At the treatment response assessment (After 6-12 cycles of treatment up to 52 weeks)
Transfusion independence (yes/no) | At the treatment response assessment (After 6-12 cycles of treatment up to 52 weeks)
General condition improvement (yes/no) | At the treatment response assessment (After 6-12 cycles of treatment up to 52 weeks)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Nancy, Nancy
  - BROSEUS, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254
- [Result] Bejar R, Stevenson K, Abdel-Wahab O, Galili N, Nilsson B, Garcia-Manero G, Kantarjian H, Raza A, Levine RL, Neuberg D, Ebert BL. Clinical effect of point mutations in myelodysplastic syndromes. N Engl J Med. 2011 Jun 30;364(26):2496-506. doi: 10.1056/NEJMoa1013343. PMID 21714648
- [Result] Chen G, Broseus J, Hergalant S, Donnart A, Chevalier C, Bolanos-Jimenez F, Gueant JL, Houlgatte R. Identification of master genes involved in liver key functions through transcriptomics and epigenomics of methyl donor deficiency in rat: relevance to nonalcoholic liver disease. Mol Nutr Food Res. 2015 Feb;59(2):293-302. doi: 10.1002/mnfr.201400483. Epub 2014 Dec 9. PMID 25380481
- [Result] Cheson BD, Greenberg PL, Bennett JM, Lowenberg B, Wijermans PW, Nimer SD, Pinto A, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Gore SD, Schiffer CA, Kantarjian H. Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia. Blood. 2006 Jul 15;108(2):419-25. doi: 10.1182/blood-2005-10-4149. Epub 2006 Apr 11. PMID 16609072
- [Result] Delhommeau F, Dupont S, Della Valle V, James C, Trannoy S, Masse A, Kosmider O, Le Couedic JP, Robert F, Alberdi A, Lecluse Y, Plo I, Dreyfus FJ, Marzac C, Casadevall N, Lacombe C, Romana SP, Dessen P, Soulier J, Viguie F, Fontenay M, Vainchenker W, Bernard OA. Mutation in TET2 in myeloid cancers. N Engl J Med. 2009 May 28;360(22):2289-301. doi: 10.1056/NEJMoa0810069. PMID 19474426
- [Result] Fandy TE, Herman JG, Kerns P, Jiemjit A, Sugar EA, Choi SH, Yang AS, Aucott T, Dauses T, Odchimar-Reissig R, Licht J, McConnell MJ, Nasrallah C, Kim MK, Zhang W, Sun Y, Murgo A, Espinoza-Delgado I, Oteiza K, Owoeye I, Silverman LR, Gore SD, Carraway HE. Early epigenetic changes and DNA damage do not predict clinical response in an overlapping schedule of 5-azacytidine and entinostat in patients with myeloid malignancies. Blood. 2009 Sep 24;114(13):2764-73. doi: 10.1182/blood-2009-02-203547. Epub 2009 Jun 22. PMID 19546476
- [Result] Greenberg PL, Tuechler H, Schanz J, Sanz G, Garcia-Manero G, Sole F, Bennett JM, Bowen D, Fenaux P, Dreyfus F, Kantarjian H, Kuendgen A, Levis A, Malcovati L, Cazzola M, Cermak J, Fonatsch C, Le Beau MM, Slovak ML, Krieger O, Luebbert M, Maciejewski J, Magalhaes SM, Miyazaki Y, Pfeilstocker M, Sekeres M, Sperr WR, Stauder R, Tauro S, Valent P, Vallespi T, van de Loosdrecht AA, Germing U, Haase D. Revised international prognostic scoring system for myelodysplastic syndromes. Blood. 2012 Sep 20;120(12):2454-65. doi: 10.1182/blood-2012-03-420489. Epub 2012 Jun 27. PMID 22740453
- [Result] Itzykson R, Kosmider O, Cluzeau T, Mansat-De Mas V, Dreyfus F, Beyne-Rauzy O, Quesnel B, Vey N, Gelsi-Boyer V, Raynaud S, Preudhomme C, Ades L, Fenaux P, Fontenay M; Groupe Francophone des Myelodysplasies (GFM). Impact of TET2 mutations on response rate to azacitidine in myelodysplastic syndromes and low blast count acute myeloid leukemias. Leukemia. 2011 Jul;25(7):1147-52. doi: 10.1038/leu.2011.71. Epub 2011 Apr 15. PMID 21494260
- [Result] Meldi K, Qin T, Buchi F, Droin N, Sotzen J, Micol JB, Selimoglu-Buet D, Masala E, Allione B, Gioia D, Poloni A, Lunghi M, Solary E, Abdel-Wahab O, Santini V, Figueroa ME. Specific molecular signatures predict decitabine response in chronic myelomonocytic leukemia. J Clin Invest. 2015 May;125(5):1857-72. doi: 10.1172/JCI78752. Epub 2015 Mar 30. PMID 25822018
- [Result] Nazha A, Narkhede M, Radivoyevitch T, Seastone DJ, Patel BJ, Gerds AT, Mukherjee S, Kalaycio M, Advani A, Przychodzen B, Carraway HE, Maciejewski JP, Sekeres MA. Incorporation of molecular data into the Revised International Prognostic Scoring System in treated patients with myelodysplastic syndromes. Leukemia. 2016 Nov;30(11):2214-2220. doi: 10.1038/leu.2016.138. Epub 2016 May 20. PMID 27311933
- [Result] Rasmussen KD, Jia G, Johansen JV, Pedersen MT, Rapin N, Bagger FO, Porse BT, Bernard OA, Christensen J, Helin K. Loss of TET2 in hematopoietic cells leads to DNA hypermethylation of active enhancers and induction of leukemogenesis. Genes Dev. 2015 May 1;29(9):910-22. doi: 10.1101/gad.260174.115. Epub 2015 Apr 17. PMID 25886910
- [Result] Santini V, Melnick A, Maciejewski JP, Duprez E, Nervi C, Cocco L, Ford KG, Mufti G. Epigenetics in focus: pathogenesis of myelodysplastic syndromes and the role of hypomethylating agents. Crit Rev Oncol Hematol. 2013 Nov;88(2):231-45. doi: 10.1016/j.critrevonc.2013.06.004. Epub 2013 Jul 7. PMID 23838480
- [Result] Sperling AS, Gibson CJ, Ebert BL. The genetics of myelodysplastic syndrome: from clonal haematopoiesis to secondary leukaemia. Nat Rev Cancer. 2017 Jan;17(1):5-19. doi: 10.1038/nrc.2016.112. Epub 2016 Nov 11. PMID 27834397